CLINICAL TRIAL: NCT04760652
Title: CBT-ENDURE: Cognitive Behavioral Therapy Following Esketamine for Major Depression and Suicidal Ideation for Relapse Prevention
Brief Title: Cognitive Behavioral Therapy Following Esketamine for Major Depression and Suicidal Ideation for Relapse Prevention
Acronym: ENDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029473; 1265736169 (Other: National Provider Identifier (NPI) #); 1R01MH125205-01 (NIH)
Record Dates: First submitted 2021-02-04; First posted 2021-02-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Depression and Suicide
Keywords: Depression; Suicide
MeSH Terms: conditions — Depression; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Esketamine:All participants will receive esketamine for MDSI (Major depression with suicidal ideation) as part of their standard care. The protocol will adhere to the FDA label for this product and the FDA-registered trials.
  CBT:Half of participants will be randomized to the CBT intervention, which will consist of an in-person and computer-based component (based on Good Days Ahead). In total, this will consist of 20 total sessions given over 16 weeks (the first 4 weeks of CBT will have sessions twice weekly; thereafter sessions will be held weekly).
  TAU only:Participants not randomized to CBT will undergo treatment as usual (TAU). These patients will undergo standard, post-hospitalization clinical treatments, which may include physician visits and psychotherapy (except for formal CBT).
Who Masked: Outcomes Assessor
Masking Description: Rater blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT Cognitive Behavioral Therapy (Active Comparator): Participants will receive CBT, which will consist of in-person and computer-based component (based on Good Days Ahead). This will consist of 20 sessions given over 16 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy CBT
- TAU Treatment As Usual (Other): Participants will undergo Treatment as usual (TAU). These patients will undergo standard, post-hospitalization clinical treatments, which many include physician visits and psychotherapy (except for formal CBT).
  Interventions: Behavioral: Cognitive Behavioral Therapy CBT

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy CBT — CBT: In-person and computer-based components (Good Days Ahead) First 4 weeks of CBT are twice weekly; thereafter weekly CBT

SUMMARY:
This is a rater-blinded, randomized controlled trial. All patients will receive esketamine for treatment of Major Depression with Suicidal Ideation (MDSI). Subjects will be randomized (1:1) to receive CBT (computer-assisted) or TAU alone following esketamine.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the feasibility and safety of performing a larger study examining the effectiveness and mechanism of action of CBT to improve the longer-term outcomes following esketamine treatment in patients hospitalized for suicidal ideation or suicide attempt.

Specific Aim 2: To evaluate the appropriateness and utility of the proposed tests of cognitive control measures in exploring the mechanisms underlying the effects on depression of esketamine and the combination of esketamine+CBT.

Specific Aim 3: To examine the efficacy of esketamine+CBT combination compared to esketamine+TAU in reducing suicidal ideation.

In August 2022, the targeted enrollment was expanded to include outpatient participants, the anticipated enrollment was increased from 60 to 100 participants as a result.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible for the study if they meet all the following criteria:

  1. Written informed consent before any study procedures are performed
  2. Meeting criteria for inpatient admission for suicidal ideation or attempt at one of the study sites
  3. Recommended by a physician for esketamine treatment
  4. Males or females ages 18 through 65 years of age
  5. Diagnosis of major depressive disorder as confirmed by the MINI (inpatient) or the HAM-D-17 (outpatient)
  6. Willing to adhere to a reliable form of contraception throughout the trial and for one month following completion of the trial (for subjects who are sexually active)
  7. In the opinion of the investigator, the patient is willing and able to comply with scheduled visits, treatment plan, and other trial procedures for the duration of the study

Exclusion Criteria:

* Participants are excluded if they meet any of the following criteria:

  1. Active substance use disorder (except tobacco) within 6 months of screening date
  2. Meets DSM-5 criteria for bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, or pervasive development disorder
  3. Dementia or other cognitive disorder or intellectual disability that would impair the subject's ability to meaningfully engage in CBT (per investigator judgment)
  4. Any other medical or psychiatric comorbidity that the investigator judges would put the participant at additional undue risk due to study participation or would impair subject's ability to participate in the study.
  5. Current or planned participation in a formal CBT program defined by the following characteristics, each session has an agenda, a homework assignment is given at each session, and the homework assignment from the previous session is reviewed at the following appointment.
  6. Previous Esketamine or ketamine treatment that did not produce a clinical response as outlined below.

     * 6 treatments with Esketamine at a dose of 56 mg or more with no clinical response
     * 6 treatments of IV ketamine at a dose between 0.4 mg/kg and 0.7mg /kg with no clinical response Patients must not have received Esketamine or ketamine treatment within the past 12 weeks of time of enrollment.
  7. The patient is pregnant or breastfeeding
  8. Unable to give informed consent
  9. Was previously enrolled/randomized into the trial
  10. Patients who have a contraindication to receiving Esketamine including any of the following:

      * aneurysmal vascular disease
      * arteriovenous malformation
      * history of intracerebral hemorrhage
      * hypersensitivity to esketamine or ketamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of performing a larger study with similar design by measuring of recruitment rates. | Recruitment rates will be assessed at 18 months.
  Feasibility will be evaluated by measures of recruitment rates measured by attaining 80% of recruitment target will be considered feasible.
To determine the feasibility of performing a larger study with similar design by measuring attrition. | Attrition will be assessed at 18 months.
  Feasibility will be evaluated by measures of attrition rates by attaining 80% of retention will of 70% of participants will be considered feasible.
Reasons for discontinuation | Discontinuation will be assessed at 18 months.
  Feasibility will be evaluated by measures of reasons for discontinuation regardless of clinical state, to Week 18 or later will be considered feasible.
To determine the safety of performing a larger study with similar design. | Safety will be assessed at 18 months.
  Safety will be evaluated by measures of the number by type of protocol deviations.
Evaluate the appropriateness of the proposed tests of cognitive control measures in exploring the mechanisms of change. | The appropriateness will be assessed at the end of study (18 months).
  Appropriateness will be evaluated by the proportion of patients who are able to complete the cognitive control assessments. As this is a feasibility study, we do not have pre-specified quantitative cutoffs.

SECONDARY OUTCOMES:
Efficacy of esketamine/CBT combination compared to esketamine/TAU in reducing the risk of suicide. | Measured at Baseline, study day 2, study day 15, study day 30, weeks 7 - 17, week 18, week 26. The primary observation will be the last observation carried forward per protocol at Week 18.
  Efficacy will be measured by the response to the MADRS (Montgomery-Asberg Depression Rating Scale). The MADRS is a 10 question assessments conducted in an interview setting.

OTHER OUTCOMES:
To evaluate the depression assessments BDI-II (Beck Depression Inventory). | BDI-II will be measured at Baseline, study day 2, study day 15, study day 30, weeks 7 - 17, week 18, week 26. The primary assessment of this outcome will be at Week 18.
  The BDI-II range of values is 0-42 and the clinical interpretation are indicated with higher scores indicating greater severity of illness.
To evaluate the depression assessments CGI (Clinical Global Impression for Severity of Suicidality). | CGI will be measured at Baseline, study day 2, study day 15, study day 30, weeks 7 - 17, week 18, week 26. The primary assessment of this outcome will be at Week 18.
  The CGI range of values is 1-5 and the clinical interpretation is indicated with higher scores indicating greater severity of illness.
To evaluate the Suicide Ideation assessments CSSRS (COLUMBIA-SUICIDE SEVERITY RATING SCALE). | The CSSRS will be measured at Baseline, study day 2, study day 15, study day 30, weeks 7 - 17, week 18, week 26. The primary assessment of this outcome will be at Week 18.
  The CSSRS range of values 0-5 and the clinical interpretation is indicated with higher score indicating greater severity.
To evaluate the BSI (Beck Scale for Suicidal Ideation). | The BSI will be measured at Baseline, study day 2, study day 15, study day 30, weeks 7 - 17, week 18, week 26. The primary assessment of this outcome will be at Week 18.
  The BSI range of values 0-63 and the clinical interpretation is indicated with higher scores indicating greater severity of illness.
To evaluate the RRS (Ruminative Responses Scale). | We will compare at Week 18 using last observation carried forward per protocol.
  RRS range of values is 22-88, with higher scores indicating greater severity.
To evaluate the SoCT (Skills of Cognitive Therapy. | We will compare at Week 18 using last observation carried forward per protocol.
  SoCT range of values is 8-40, with higher scores indicating greater mastery of CBT.
To evaluate CTAS (Computer-Assisted Cognitive-Behavior Therapy for Depression). | We will compare at Week 18 using last observation carried forward per protocol.
  CTAS range of values is 0-40, with higher scores indicating greater knowledge of CBT.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Wilkinson, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - UAB Medicine | Heersink School of Medicine, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No